CLINICAL TRIAL: NCT04309448
Title: Augmenting Reactive Stepping With Functional Electrical Stimulation for Individuals Living With Incomplete Spinal Cord Injury
Brief Title: Augmenting Reactive Stepping With FES After SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-5462
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perturbation-based balance training with FES (Experimental)
  Interventions: Behavioral: Perturbation-based balance training with functional electrical stimulation

INTERVENTIONS:
Behavioral: Perturbation-based balance training with functional electrical stimulation — The PBT program will consist of repetitive practice of reactive stepping for one hour. The participants will be equipped with the Odstock 2-Channel stimulator on one or both sides depending on their deficits. One channel of stimulation may be applied to the common fibular nerve to elicit a flexor withdraw reflex and elicit a step. The second channel of stimulation may be applied to the quadriceps muscles to assist with the supporting phase of the reactive step, as required. Participants will experience about 60 perturbations per session during balance exercises. To create a perturbation, the researcher will apply unexpected pushes or pulls to a safety harness around the participant's trunk. Throughout the hour-long session, participants will complete challenging balance tasks, customized to their ability level, during standing and walking. The training will be supervised by a licensed physiotherapist and administered by a licensed physiotherapist or registered kinesiologist.

SUMMARY:
Up to 25 individuals living with chronic incomplete spinal cord injury (iSCI) who can stand but have limited ability to elicit a step without physical assistance or upper limb (U/L) support will be recruited for this study. The first objective of the study will aim to investigate the orthotic effect (i.e., immediate effect) of FES on the reactive stepping response. The second objective is to investigate the therapeutic effect of a novel balance intervention, perturbation-based balance training (PBT) combined with FES (i.e., PBT+FES) on reactive stepping ability, measures of postural sway during quiet standing (i.e., biomechanical measures), and scores on clinical measures of balance and walking.

ELIGIBILITY:
Inclusion Criteria:

1. have a motor incomplete SCI (i.e., AIS grade C or D) that is non-progressive;
2. be at least one year post-injury (i.e., chronic injury);
3. ≥ 18 years old;
4. be able to stand independently for 60 sec;
5. unable to take a step bilaterally without physical assistance or upper extremity support;
6. able to understand spoken English;
7. free of any other condition besides SCI that significantly affects walking or balance (e.g., no vestibular disorder, significant vision loss, stroke);
8. be able to provide informed, written consent.

Exclusion Criteria:

1. Contraindications for EMS. Electrical stimulation will not be used if:

   * it will be applied to areas where it could cause malfunction of electronic devices, including cardiac pacemakers;
   * a woman is pregnant;
   * the applied region has known or suspected malignancy;
   * the person has active deep vein thrombosis or thrombophlebitis;
   * there are active bleeding tissues, or the person has untreated hemorrhagic disorders;
   * there are infected tissues, tuberculosis, or wounds with underlying osteomyelitis;
   * tissues have been radiated in the past six months;
   * there are damaged skin areas or at-risk skin areas that would result in uneven conduction of current;
2. severe spasticity is present in the legs;
3. the person has contractures in the lower limbs that prevent achieving a neutral hip and ankle position, or extended knee;
4. there is a history of prior lower limbs fragility fracture;
5. the leg muscles are unresponsive to electrical stimulation (i.e., peripheral nerve damage in the legs).
6. Pressure sores on pelvis or trunk, where safety harness will be donned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Lean-and-release test | Up to 7 weeks
  Test of reactive stepping and balance in the forward direction
Biomechanical measures of postural control | Up to 7 weeks
  Measurement of centre of pressure during quiet standing

SECONDARY OUTCOMES:
Mini-Balance Evaluation Systems Test | Up to 7 weeks
  Assesses four balance control systems
Activities-specific Balance Confidence Scale | Up to 7 weeks
  Assesses balance efficacy
Gait parameters | Up to 7 weeks
  Step length (cm), gait speed (m/s), double support time (%)
Falls Efficacy Scale International | Up to 7 weeks
  Assesses the degree of concern about fear of falling
Semi-structured interview | 3 months post
  Queries the participants' perceived challenges and benefits of the PBT+FES program

CONTACTS AND LOCATIONS:
Locations (1):
- Lyndhurst Centre, Toronto Rehabilitation Institute-UHN, Toronto, Ontario, Canada